CLINICAL TRIAL: NCT06387342
Title: CF102-222PC: A Phase 2 Open-Label Study of the Safety and Activity of Namodenoson in the Treatment of Advanced Pancreatic Adenocarcinoma
Brief Title: Namodenoson Treatment of Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF102-222PC
Record Dates: First submitted 2024-04-15; First posted 2024-04-29 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Namodenoson 25 mg (Experimental): namodenoson capsule, 25 mg, administered orally, twice daily for consecutive 28-day cycles
  Interventions: Drug: Namodenoson 25mg

INTERVENTIONS:
Drug: Namodenoson 25mg — oral capsule
  Other Names: CF102

SUMMARY:
This is an open-label trial in patients with advanced pancreatic cancer. The trial will evaluate the safety, clinical activity, and pharmacokinetics of the study drug, namodenoson, in this group of patients.

DETAILED DESCRIPTION:
All patients will receive the study drug twice daily. The study drug is given as a capsule, orally (by mouth). Patients will be monitored regularly for safety. Tumor imaging will be performed approximately every two months. Patients can decide to stop the treatment with study drug at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Histologically or cytologically confirmed pancreatic adenocarcinoma, or clinically diagnosed based upon scan results and a serum Cancer Antigen 19-9 value >1000 U/mL on at least 1 occasion.
3. Pancreatic adenocarcinoma is advanced (i.e., treatment-refractory or metastatic) and no standard therapies are expected to be curative.
4. Pancreatic adenocarcinoma has progressed on at least 1 prior systemic treatment regimen, or the patient refuses standard treatment.
5. Prior pancreatic adenocarcinoma treatment was discontinued for at least 14 days prior to the Baseline Visit.
6. Measurable or evaluable disease by RECIST v1.1.
7. Patients with a history of treated central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria: disease outside the CNS is present; there is no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study; and there is no history of intracranial hemorrhage or spinal cord hemorrhage.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of ≤ 2.
9. The following laboratory values must be documented prior to the first dose of study drug:

   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelet count ≥50 × 109/L
   * Creatinine clearance ≥50 mL/min (estimated glomerular filtration rate by the Cockcroft-Gault) or serum creatinine ≤2.0 mg/dL
   * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) ≤10X the upper limit of normal
   * Total bilirubin ≤10 mg/dL
   * Serum albumin ≥2.0 g/dL.
10. Life expectancy of ≥8 weeks.
11. For women of childbearing potential, negative serum pregnancy test result.
12. Provide written informed consent to participate.
13. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other trial-related procedures

Exclusion Criteria:

1. Receipt of systemic cancer therapy within 14 days prior to the Baseline Visit or concurrently during the trial.
2. Persistent toxicity ≥Grade 2 from previous cancer therapy, with the exceptions of alopecia and Grade 3 peripheral neuropathy.
3. Major surgery or radiation therapy within 14 days prior to the Baseline Visit.
4. Use of any investigational agent within the shorter of 4 weeks or 5 half-lives prior to the Baseline Visit.
5. Concomitant use of P-glycoprotein (P-gp)/breast cancer resistance protein (BCRP) inhibitors and/or substrates with a narrow therapeutic index unless the medication can be taken at least 3 hours before or after taking the investigational product.
6. Unable to swallow orally administered medication or presence of a gastrointestinal disorder likely to interfere with absorption of the study medication.
7. Uncontrolled or clinically unstable thyroid disease, per judgment of the Principal Investigator.
8. Active bacterial, viral, or fungal infection requiring systemic therapy or operative or radiological intervention.
9. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness or other immunodeficiency.
10. Active second primary malignancy (other than pancreatic adenocarcinoma) requiring treatment.
11. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4).
12. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 1 month prior to initiation of study drug.
13. History of, or ongoing, cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the corrected QT interval (QTc) (Fridericia) interval to >470 msec [mean of triplicate electrocardiogram measurements] (patients with bundle branch block or a cardiac pacemaker will not be excluded for QTc reasons).
14. Pregnant or lactating female.
15. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Investigator, are effective and adequate for the patient's circumstances while on study drug and for at least 1 month thereafter.
16. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 1 month afterward.
17. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with trial participation or study drug administration; may interfere with the informed consent process and/or with compliance with the requirements of the trial; or may interfere with the interpretation of trial results and, in the Investigator's opinion, would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Every 2 weeks, assessed up to 1 year
  Assessments of adverse events (AEs) will include characterization of type, incidence, severity (graded by CTCAE v5.0), seriousness, and relationship to treatment.
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Change from baseline | Every 2 weeks, assessed up to 1 year
  Eastern Cooperative Oncology Group (ECOG) Performance Status (PS), which is a scale of functioning, from 0 (normal activity) to 5 (death)

SECONDARY OUTCOMES:
Objective response rate | Every 8 weeks, assessed up to 1 year
  clinical activity measure of objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), measured by computed tomography (CT) scan, positron emission tomography (PET) CT, and/or magnetic resonance imaging (MRI)
Progression free survival | Every 8 weeks, assessed up to 1 year
  clinical activity measure of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), measured by computed tomography (CT) scan, positron emission tomography (PET) CT, and/or magnetic resonance imaging (MRI)
Disease control rate | Every 8 weeks, assessed up to 1 year
  clinical activity measure of disease control rate (DCR)
Duration of response | Every 8 weeks, assessed up to 1 year
  clinical activity measure of duration of response (DoR), defined as the time from first response to disease progression or death from any cause, whichever occurs first
Overall survival | Every 8 weeks, assessed up to 1 year
  clinical activity measure of overall survival (OS), including death from any cause

OTHER OUTCOMES:
Quality of Life evaluation with EORTC QLQ-C30 | Every 4 weeks, assessed up to 1 year
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30), in which summary scores range from 0 to 100, with higher scores indicating better health-related quality of life
Quality of Life evaluation with EORTC QLQ-PAN26 | Every 4 weeks, assessed up to 1 year
  European Organization for Research and Treatment of Cancer Quality of Life pancreatic adenocarcinoma-specific module, the EORTC QLQ-PAN26, in which summary scores range from 0 to 100, with higher scores indicating better health-related quality of life
Pharmacokinetics of namodenoson: Cmax | Cycle 1, day 1 (each cycle is 28 days); Cycle 1, day 15, and Cycle 2, day 1
  Maximum plasma concentration of namodenoson
Pharmacokinetics of namodenoson: Cmin | Cycle 1, day 1 (each cycle is 28 days); Cycle 1, day 15, and Cycle 2, day 1
  Minimum plasma concentration of namodenoson
Pharmacokinetics of namodenoson: AUC(0-12) | Cycle 1, day 1 (each cycle is 28 days); Cycle 1, day 15, and Cycle 2, day 1
  Area under the curve of namodenoson plasma exposure from 0-12 hours post-dose
Cancer antigen 19-9 (CA 19-9) | Every 4 weeks, assessed up to 1 year
  Change from baseline in Cancer antigen 19-9 (CA 19-9) biomarker during treatment
Carcinoembryonic Antigen (CEA) | Every 4 weeks, assessed up to 1 year
  Change from baseline in Carcinoembryonic Antigen (CEA) biomarker during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma; Salomon M Stemmer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center Institute of Oncology, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modi S, Kir D, Banerjee S, Saluja A. Control of Apoptosis in Treatment and Biology of Pancreatic Cancer. J Cell Biochem. 2016 Feb;117(2):279-88. doi: 10.1002/jcb.25284. PMID 26206252
- [Background] Mazziotta C, Rotondo JC, Lanzillotti C, Campione G, Martini F, Tognon M. Cancer biology and molecular genetics of A3 adenosine receptor. Oncogene. 2022 Jan;41(3):301-308. doi: 10.1038/s41388-021-02090-z. Epub 2021 Nov 8. PMID 34750517
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Itzhak I, Bareket-Samish A, Fishman P. Namodenoson Inhibits the Growth of Pancreatic Carcinoma via Deregulation of the Wnt/beta-catenin, NF-kappaB, and RAS Signaling Pathways. Biomolecules. 2023 Oct 27;13(11):1584. doi: 10.3390/biom13111584. PMID 38002266
- [Background] Li L, Mo FK, Chan SL, Hui EP, Tang NS, Koh J, Leung LK, Poon AN, Hui J, Chu CM, Lee KF, Ma BB, Lai PB, Chan AT, Yu SC, Yeo W. Prognostic values of EORTC QLQ-C30 and QLQ-HCC18 index-scores in patients with hepatocellular carcinoma - clinical application of health-related quality-of-life data. BMC Cancer. 2017 Jan 4;17(1):8. doi: 10.1186/s12885-016-2995-5. PMID 28052758
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- See also: American Heart Association Classes of Heart Failure. www.heart.org. — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure